CLINICAL TRIAL: NCT03144544
Title: Incidences of Non-physiologically Complex Surgical Procedures Performed in Children and Their Similarity of Distribution Between Pediatric Specialist Hospitals and Other Hospitals Performing Pediatric Surgery
Brief Title: Physiological Complexity of Pediatric Surgery Between Types of Hospitals
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, James O'Leary, Staff Anesthesiologist, The Hospital for Sick Children
Other Study IDs: 1000053805
Record Dates: First submitted 2017-05-04; First posted 2017-05-09 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Health Services
Keywords: Similarity; Diversity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric specialist hospitals: Free-standing hospitals providing tertiary pediatric referral services and performing pediatric surgical procedures
  Interventions: Procedure: Pediatric surgical procedures
- Non-pediatric specialist hospitals: Other hospitals performing pediatric surgical procedures
  Interventions: Procedure: Pediatric surgical procedures

INTERVENTIONS:
Procedure: Pediatric surgical procedures — Eligible surgical procedures were identified using Canadian Classification of Health Interventions (CCI) therapeutic intervention codes.

SUMMARY:
When considered from a provincial perspective, quantification of surgical procedures undertaken by different hospitals and healthcare networks is necessary for informing resource allocation and modelling of healthcare services. The investigators hypothesized that i) non-physiologically complex surgical procedures would account for most (>1/2) of pediatric surgical procedures performed at both pediatric specialist hospitals and the other hospitals performing pediatric surgery, ii) surgical discharges for non-physiologically complex surgical procedures would account for most (>1/2) in-hospital bed nights among pediatric surgical admissions at both pediatric specialist hospitals and the other hospitals performing pediatric surgery, and iii) the relative distributions of non-physiologically complex surgical procedures, but not physiologically complex procedures, would be at least moderately similar between pediatric specialist hospitals and the other hospitals performing pediatric surgery. To test these 3 hypotheses, the specific objectives of this study were to estimate i) the proportion (primary outcome) of non-physiologically complex pediatric surgical procedures, and ii) the similarity and diversity (secondary outcomes) of non-physiologically and physiologically complex surgical procedures between the pediatric specialist hospitals and the other hospitals performing pediatric surgery in Ontario, Canada.

ELIGIBILITY:
Inclusion Criteria:

* surgical procedures for individuals aged greater than 27 days and less than 18 years

Exclusion Criteria:

* newborns (0 to 27 days of age)
* records lacking a patient identifier or age
* non-surgical healthcare interventions

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric surgical procedures
Sampling Method: Non-Probability Sample
Enrollment: 830830 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2016-10-27 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of non-physiologically complex surgery | April 1, 2007 to March 31, 2015
  The proportion of non-physiologically complex pediatric surgical procedures

SECONDARY OUTCOMES:
Similarity | April 1, 2007 to March 31, 2015
  Similarity of different types of pediatric surgical procedures performed between hospitals was assessed using Yue and Clayton's index
Diversity | April 1, 2007 to March 31, 2015
  Effective number of common procedures

CONTACTS AND LOCATIONS:
Overall Officials: James D O'Leary, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All relevant data are within the paper.

REFERENCES:
- [Derived] O'Leary JD, Dexter F, Faraoni D, Crawford MW. Incidence of non-physiologically complex surgical procedures performed in children: an Ontario population-based study of health administrative data. Can J Anaesth. 2018 Jan;65(1):23-33. doi: 10.1007/s12630-017-0993-y. Epub 2017 Nov 17. PMID 29150783